CLINICAL TRIAL: NCT03659305
Title: Double-blind Randomized Comparative, in Parallel Groups, Clinical Study of Pharmacokinetics and Safety of Drugs RPH-001 (JSC R-Pharm, Russia) and Avastin® (F. Hoffmann-La Roche Ltd, Switzerland) in Single Intravenous Administration in Healthy Volunteers
Brief Title: Pharmacokinetic Equivalence and Safety Study of RPH-001 and Avastin®
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: R-Pharm (Industry)
Collaborators: Almedis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: СL01011063
Record Dates: First submitted 2018-09-03; First posted 2018-09-06 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: Bevacizumab; oncology; VEGF receptor
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPH-001 (Experimental): Humanized recombinant monoclonal anti-VEGF antibody. 5 mg/kg single intravenous infusion (for no less than 90 minutes)
  Interventions: Biological: RPH-001
- Avastin (Active Comparator): Humanized recombinant monoclonal anti-VEGF antibody. 5 mg/kg single intravenous infusion (for no less than 90 minutes)
  Interventions: Biological: Avastin

INTERVENTIONS:
Biological: RPH-001 — Concentrate for preparation solution for infusion in ampules, 25 mg/mL
  Other Names: Bevacizumab
  Arms: RPH-001
Biological: Avastin — Concentrate for preparation solution for infusion in ampules, 25 mg/mL
  Other Names: Bevacizumab
  Arms: Avastin

SUMMARY:
The purpose of this study is to confirm pharmacokinetic equivalence and compare clinical safety profile of RPH-001 and Avastin®.

DETAILED DESCRIPTION:
The study will be conducted in one specialized clinical site in Russia. It is planned to randomize 80 healthy male volunteers in this study. After screening period, not exceeding 15 days, all eligible subjects will be hospitalized to the site and randomized to receive RPH-001 or Avastin in 1:1 ratio. After a single-dose of investigational drugs administration subjects will remain under the observation in clinical site for 8 days and then will be discharged. The out-patient follow up period will include at least 8 scheduled subject's visits to the site. The study will consider completed for each subject at Day 100 visit after all clinical study procedures completion.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signed informed consent form prior to any research procedure.
* Body Mass Index (BMI) between 18,5 and 30 kg/m^2, inclusively, and body mass between 60 and 100 kg, inclusively.
* Verified diagnosis "Healthy" according to standard clinical, laboratory and instrumental methods of examination, namely haemodynamic parameters within normal limits: systolic blood pressure in the range of 100 - 130 mm Hg inclusive, diastolic blood pressure in the range of 60 - 90 mm Hg inclusive, heart rate is 60-90 beats/minute inclusive (according to the physical examination); the absence of deviations from the norm in the results of laboratory and instrumental methods of examination, including ECG (normal standard electrocardiogram in 12 leads after 10 minutes of rest in the supine position should meet the following parameters: 120ms < PR < 200 ms, QRS<120 ms, QTc ≤ 430 ms).
* The ability of volunteer, according to the investigator, to comply with the Protocol procedures.
* The willingness of the volunteer and his sexual partner with the preserved reproductive function to use reliable methods of contraception from the day of hospitalization (Day -1) until the end of the follow-up period (Day 100). This requirement does not apply to participants who underwent surgical sterilization. Reliable methods of contraception suggest the use of the 1-st barrier method in combination with one of the following: spermicide, intrauterine device/oral contraceptives in the sexual partner. Willingness to refuse sperm donation during the period of drug taking and until the end of the follow-up period (completion of the visit Day 100).

Exclusion Criteria:

* Chronic disease of cardiovascular, bronchopulmonary, neuroendocrine systems, as well as diseases of gastrointestinal tract, kidneys, blood and autoimmune diseases in the past history.
* Acute infections less than 4 weeks prior to the signing inform consent.
* The presence of documented history of malignant diseases.
* Mental illness and other conditions that may affect the volunteer's ability to follow the study protocol.
* Blood and/or plasma donation in excess of 450 mL within 60 days prior to the signing of informed consent and planned blood and/or plasma donation before the end of the study (completion of the visit Day 100).
* Any prior use of anti-VEGF-antibodies or any other drug targeted at the VEGF receptor, in particular Avastin or its biosimilar.
* The presence of anaphylaxis in the past history to any biological drug.
* Extensive surgical procedures including appendectomy in the last 12 weeks prior to the signing of the informed consent.
* History of drug or alcohol dependence - regular intake of more than 10 units of alcohol per week (1 unit of alcohol is equal to 500 mL of beer, 200 mL of wine or 50 mL of alcohol).
* Smoking more than 5 cigarettes a day or using an equivalent amount of tobacco, inability to stop smoking during the study.
* The use of any drugs (including drugs based on St John's Wort, with the exception of drugs used as topical application, without systemic absorption) for 14 days or for an interval of time equal to 6 half-life prior to the signing of the informed consent (depending on what time interval is longer); any vaccination within the last 28 days prior to the signing of the informed consent; the use of any biological drug (antibody or its derivative) within 4 months prior to the signing of the informed consent.
* Participation in any clinical trials of medicines less than 90 calendar days prior to the signing of the informed consent.
* Previous participation in the study of drug RPH-001.
* Any volunteer who is an investigator or co-investigator, laboratory assistant, pharmacist, research coordinator or other employee directly involved in the conduct of this study.
* A positive result of any of the following tests: hepatitis B surface antigen (HBs Ag), hepatitis C antibodies (anti-HCV), antibodies to human immunodeficiency virus 1 and 2 (anti-HIV1 and anti-HIV2), blood test for syphilis at the Screening visit.
* Positive urine test result for drugs on Screening visit and visit Day -1 (cannabis, amphetamines, methamphetamine, cocaine, morphine, barbiturates, benzodiazepines).
* Positive test result for alcohol on Screening visit and visit Day -1.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2019-01-26 (Actual); Study Completion 2019-01-26 (Actual)

PRIMARY OUTCOMES:
Cmax | 30 minutes before and 90 minutes after the start of investigational product infusion, 4, 24, 48, 96, 168, 336, 504, 672, 1008, 1344, 1512,1680 and 2376 hours after the start of investigational product infusion
  Maximum concentration of investigational drug achieved during sampling
AUC(0-t) | 30 minutes before and 90 minutes after the start of investigational product infusion, 4, 24, 48, 96, 168, 336, 504, 672, 1008, 1344, 1512,1680 and 2376 hours after the start of investigational product infusion
  Area Under the Concentration-time curve from time 0 to the time of the last sample with measurable concentration
AUC(0-∞) | 30 minutes before and 90 minutes after the start of investigational product infusion, 4, 24, 48, 96, 168, 336, 504, 672, 1008, 1344, 1512,1680 and 2376 hours after the start of investigational product infusion
  Area Under the Concentration-time curve from time 0 extrapolated to infinite time

SECONDARY OUTCOMES:
tmax | 30 minutes before and 90 minutes after the start of investigational product infusion, 4, 24, 48, 96, 168, 336, 504, 672, 1008, 1344, 1512,1680 and 2376 hours after the start of investigational product infusion
  Time at which Cmax is attained
t1/2 | 30 minutes before and 90 minutes after the start of investigational product infusion, 4, 24, 48, 96, 168, 336, 504, 672, 1008, 1344, 1512,1680 and 2376 hours after after the start of investigational product infusion
  The terminal half-life
λz | 30 minutes before and 90 minutes after the start of investigational product infusion, 4, 24, 48, 96, 168, 336, 504, 672, 1008, 1344, 1512,1680 and 2376 hours after the start of investigational product infusion
  Elimination rate constant
Vz | 30 minutes before and 90 minutes after the start of investigational product infusion, 4, 24, 48, 96, 168, 336, 504, 672, 1008, 1344, 1512,1680 and 2376 hours after the start of investigational product infusion
  Apparent Volume of Distribution

OTHER OUTCOMES:
Immunogenicity | 30 minutes before and 336, 672, 1344, 1680 and 2376 hours after the start of investigational product infusion
  Anti-drug-antibodies (ADA), Neutralizing antibodies (NAb)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — R-Pharm
Locations (1):
- SBHI Krasnogorskaya City Hospital #1, Krasnogorsk, Russia